CLINICAL TRIAL: NCT01175148
Title: Phase II Study Evaluating the Safety and Efficacy of Atorvastatin for the Prophylaxis of Acute Graft-versus-host Disease in Patients Undergoing Matched Sibling Hematopoietic Stem Cell Transplantation
Brief Title: Atorvastatin for the Prophylaxis of Acute GVHD in Patients Undergoing Matched Sibling Allogeneic Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WVU11010
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Graft vs Host Disease
Keywords: HSCT; HPC; HCT; BMT; lipitor; atorvastatin; HMG-CoA Reductase Inhibitor; Hematopoietic stem cell transplant; allogeneic transplant; GVHD; graft-versus-host-disease; Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recipient - Atorvastatin to prevent GVHD (Experimental): Atorvastatin calcium (Lipitor) will be administered at dose of 40mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning. Patients will receive atorvastatin until +180 days or development of grade 2 GVHD. This is the experimental arm for outcome measures.
  Interventions: Drug: Atorvastatin calcium (Lipitor)
- Donor - Atorvastatin conditioning for donors (Other): Sibling donors will start taking Atorvastatin calcium (Lipitor) orally at 40mg once daily between 14-28 days before the anticipated first day of apheresis or bone marrow harvest.
  Interventions: Drug: Atorvastatin calcium (Lipitor)

INTERVENTIONS:
Drug: Atorvastatin calcium (Lipitor) — 40 mg PO daily
  Other Names: Lipitor

SUMMARY:
Atorvastatin for prevention of acute GVHD

DETAILED DESCRIPTION:
This is a phase II study of atorvastatin for the prophylaxis of acute GVHD in patients undergoing matched-sibling allogeneic HSCT. This study will explore a two-pronged acute GVHD prophylaxis strategy, consisting of pre-treating consenting sibling donors with atorvastatin before stem cell collection, followed by the addition of atorvastatin to methotrexate/tacrolimus-based GVHD prophylaxis.

ELIGIBILITY:
DONOR ELIGIBILITY CRITERIA:

1. Donors must be ≥18 years of age, and willing/able to provide informed consent.
2. Female donors of child-bearing potential should have a negative pregnancy test, and must be not be breast feeding.
3. Adequate hepatic function with bilirubin, AST and ALT < 2.5 x upper limit of normal.
4. Adequate renal function as defined by a serum creatinine clearance of ≥ 40% of normal calculated by Cockcroft-Gault equation.
5. Adequate cardiac function as per institutional guidelines.
6. Donors with positive HIV serologies are not eligible.
7. No clinical evidence of uncontrolled active bacterial, viral or fungal infection at the time of stem cell mobilization.
8. Donors must have a Karnofsky performance score of ≥60.
9. Donors with history of intolerance or allergic reactions with atorvastatin will not be eligible. Hypersensitivity to any component of atorvastatin.
10. Method of stem-cell collection from the sibling donor will be at the discretion of the treating physician. Although it is anticipated that majority of sibling donors will undergo G-CSF induced stem cell mobilization; however donors undergoing bone marrow harvest or stem cell mobilization with experimental agents (e.g. plerixafor) will remain eligible for the study.

PATIENT ELIGIBILITY CRITERIA:

1. Patients with a history of a hematological malignancy or bone marrow failure syndrome suitable for matched sibling allogeneic stem cell transplantation in the opinion of treating transplant physician.
2. Patients aged 18-75 years of age are eligible. Patients with age > 18 and ≤ 50 years will be eligible for myeloablative conditioning (MAC), while patients > 50 years of age, or those with previous history of autologous transplantation, high hematopoietic cell transplant comorbidity index (HCT-CI) score (>2), and baseline diagnosis of hodgkin's lymphoma, chronic lymphocytic leukemia and follicular lymphoma will be suitable for reduced intensity conditioning (RIC) transplantation (however intensity of conditioning regimen will remain at the discretion of treating physician).
3. All patients must have at least one suitable HLA-matched sibling donor according to transplant center's guidelines (for selection of appropriate sibling donor).
4. Patient must provide informed consent.
5. Left ventricular ejection fraction > 40%. No uncontrolled arrhythmias or uncontrolled New York Heart Association class III-IV heart failure.
6. Bilirubin <2mg/dl and AST and ALT < 3 x normal; and absence of hepatic cirrhosis.
7. Adequate renal function as defined by a serum creatinine clearance of ≥ 40% of normal calculated by Cockcroft-Gault equation.
8. DLCO (diffusion capacity; corrected for hemoglobin) ≥ 50% of predicted.
9. Karnofsky performance status > 70.
10. A negative pregnancy test will be required for all women of child bearing potential. Breast feeding is not permitted.
11. Patients with positive HIV serology are not eligible.
12. No evidence of active uncontrolled bacterial, viral or fungal infection at the time of transplant conditioning.
13. Patients with history of intolerance or allergic reactions with atorvastatin will not be eligible.
14. Patients who have previously been taking atorvastatin or any other statin drug will be eligible as long as there is no contraindication to switch to atorvastatin (40mg/day) in the opinion of the treating physician.
15. Patients undergoing a T-cell depleted allogeneic transplantation will not be eligible.
16. Patients receiving conditioning regimens containing antithymocyte globulin, and/or campath will not be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hamadani, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Hamadani M, Awan FT, Devine SM. The impact of HMG-CoA reductase inhibition on the incidence and severity of graft-versus-host disease in patients with acute leukemia undergoing allogeneic transplantation. Blood. 2008 Apr 1;111(7):3901-2. doi: 10.1182/blood-2008-01-132050. No abstract available. PMID 18362217
- [Background] Zeiser R, Youssef S, Baker J, Kambham N, Steinman L, Negrin RS. Preemptive HMG-CoA reductase inhibition provides graft-versus-host disease protection by Th-2 polarization while sparing graft-versus-leukemia activity. Blood. 2007 Dec 15;110(13):4588-98. doi: 10.1182/blood-2007-08-106005. Epub 2007 Sep 7. PMID 17827390

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipient Arm: Atorvastatin will be administered at dose of 40mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning. Patients will receive atorvastatin until +180 days or development of grade 2 GVHD.
  Atorvastatin calcium (Lipitor): 40 mg PO daily
- Donor Arm: Sibling donors will start taking atorvastatin orally at 40mg once daily between 14-28 days before the anticipated first day of apheresis or bone marrow harvest.
Period: Overall Study
Arm/Group | Recipient Arm | Donor Arm
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recipient Arm | Donor Arm | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Number; unit: participants]
  18-49 | 10 | 11 | 21
  50--69 | 19 | 17 | 36
  70-80 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Cummalative Incidence of Grade 2 to 4 Acute Graft vs Host Diesease (GVHD) at Day 100 Post Transplant in HSCT Recipients
Description: Cummalative incidence of grade 2 to 4 acute Graft vs Host Diesease (GVHD) at day 100 post transplant will be will be histologically confirmed and graded in Hematopoietic Stem Cell Transplantation Recipients
Time Frame: 100 days post transplant
Population: Only the Recipients were analyzed for the outcome measurements.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Recipient Arm - Experimental: Atorvastatin will be administered at dose of 40mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning. Patients will receive atorvastatin until +180 days or development of grade 2 GVHD.
  Atorvastatin calcium (Lipitor): 40 mg PO daily
Arm/Group | Recipient Arm - Experimental
Number analyzed (Participants) | 30
percentage of participants | 3.3 [0.2 to 14.8]
Statistical Analysis 1: Comparison: Recipient Arm - Experimental; The study used a minimax Simon two-stage design to test the null hypothesis Ho: P > 0.35 versus the alternative H1: < 0.15, where P is the probability of grade 2 to 4 acute GVHD at day + 100; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = .15

ADVERSE EVENTS:
Time Frame: 2 years from study enrollment
Arm/Group | Recipient Arm - Experimental | Donor Arm
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 8/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recipient Arm - Experimental (N=30) | Donor Arm (N=30)
Myalgias (Musculoskeletal and connective tissue disorders) | 3 | 0
Ankle Edema (Blood and lymphatic system disorders) | 1 | 0
Fatigue (Nervous system disorders) | 1 | 0
Liver Function Tests (Hepatobiliary disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No